CLINICAL TRIAL: NCT00391560
Title: Phase II Study of Perifosine in Patients With Refractory and Relapsed Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 217
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2012-02

CONDITIONS: Leukemia
Keywords: refractory leukemia
MeSH Terms: conditions — Leukemia | interventions — perifosine

STUDY DESIGN:
Intervention Model Description: Single treatment arm. Two disease related analyses groups, i.e.: Group 1: AML, MDS, CML-BP non-lymphoid, CMML, Agnogenic Myeloid Metaplasia (AMM); Group 2: CLL, ALL, CML-BP lymphoid
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 on Perifosine (Experimental): Patients with AML, MDS, CML-BP non-lymphoid, CMML, or Agnogenic Myeloid Metaplasia (AMM).
  After a one-time loading dose of 600 mg (150 mg x 4 at least 4 hours apart) during the first cycle, perifosine will be given orally at 100 mg once a day continuously. Cycles are 28 days in length.
  Intra-patient dose escalation for the maintenance dose to 150 mg daily will be done in the second cycle if no non-hematological toxicities beyond grade 0-1 occurred during the first cycle are observed.
  Interventions: Drug: perifosine
- Group 2 on Perifosine (Experimental): Patients with CLL, ALL, or CML-BP lymphoid. After a one-time loading dose of 600 mg (150 mg x 4 at least 4 hours apart) during the first cycle, perifosine will be given orally at 100 mg once a day continuously. Cycles are 28 days in length.
  Intra-patient dose escalation for the maintenance dose to 150 mg daily will be done in the second cycle if no non-hematological toxicities beyond grade 0-1 occurred during the first cycle are observed.
  Interventions: Drug: perifosine

INTERVENTIONS:
Drug: perifosine — Identical intervention in both arms.
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a Phase II trial designed to determine the efficacy and safety of perifosine in patients with leukemia who develop progressive disease or recurrence while receiving therapy.

DETAILED DESCRIPTION:
This is a Phase II study of perifosine in patients with refractory and relapsed leukemia. After a one time loading dose of 600 mg (150 mg x 4 at least 4 hours apart) during the first cycle, perifosine will be given orally at 100 mg once a day continuously. Cycles are 28 days in length. Intra-patient dose escalation for the maintenance dose to 150 mg daily will be done in the second cycle if no non-hematological toxicities beyond grade 0-1 occurred during the first cycle are observed.

Patients will be assessed for efficacy at the end of each 28 day cycle of therapy, +/- 7 days. Complete remissions, partial remissions and hematological improvements of any kind will be counted towards an objective response for all diseases.

A maximum total of 74 patients will be enrolled on the study, all of them assigned to the same experimental treatment scheme (arm) described above.

A maximum total of 37 evaluable patients will be entered in each of two diagnostic groups, which are being distinguished due to different anticipated rates of accrual. Group 1: AML, MDS, CML-BP non-lymphoid, CMML, Agnogenic Myeloid Metaplasia (AMM); Group 2: CLL, ALL, CML-BP lymphoid.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable remission. Patients with poor-risk myelodysplasia (MDS) [i.e. refractory anemia with excess blasts (RAEB-1 or RAEB-2) by WHO classification] and chronic myelomonocytic leukemia (CMML) are also candidates for this protocol. Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML) by WHO classification, acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Patients with agnogenic myeloid metaplasia (AMM) are also eligible.
* ECOG performance status of 0-2
* Sexually active men and women who are not surgically sterile or post menopausal must use acceptable contraceptive methods (physician will discuss acceptable methods) during the time on study and for 4 weeks following the completion of treatment. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this trial.
* In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least five half-lives for noncytotoxic agents. Persistent chronic toxicities from prior chemotherapy must not be greater than grade 1.
* Patients must have the following clinical laboratory values:

  * Serum creatinine: <= 2.0 mg/dl
  * Total bilirubin: <=1.5x the upper limit of normal unless considered due to Gilbert's syndrome
  * Alanine aminotransferase (ALT), or aspartate aminotransferase (AST): <= 3x the upper limit of normal unless considered due to organ leukemic involvement
* Must be able and willing to give written informed consent
* Age equal to or greater than 18 years

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure
* Patients with a history of severe hyper-reactive airway system (e.g. active asthma, COPD)
* Patients receiving any other standard or investigational treatment for their hematologic malignancy
* Pregnant and nursing patients are excluded because the effects of perifosine on a fetus or nursing child are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (CR + PR) | Every 4 weeks
  All patients included in the study must be assessed for response to treatment, unless there are major protocol treatment deviations or they are ineligible.
  Even a 5% response rate would be of interest for this agent, given the different nature and mechanism of action of this compound.

SECONDARY OUTCOMES:
Time to Tumor Progression | Every 4 weeks
  "Time to Progression" is defined as the period of time from the date of first study drug administration to the date that the patient is withdrawn because of clinical or radiographic progressive disease or death from any cause.
Hematologic Improvement | Every 4 weeks
  Hematological improvements of any kind will be counted towards an objective response for all diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Giles, MD, Study Chair — M.D. Anderson Cancer Center